CLINICAL TRIAL: NCT05000827
Title: Multi-institutional Evaluation of the Cost-effectiveness of PSMA-PET/CT for the Detection of Pelvic Lymph Node Invasion in Newly Diagnosed Prostate Cancer Patients
Brief Title: Dutch National Randomized Study: PSMA-PET/CT As a Triage Tool for Pelvic Lymph Node Dissection in Prostatectomy Patients
Acronym: PSMA-SELECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canisius-Wilhelmina Hospital (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL76042.091.21; 2021-8189 (Registry Identifier: CMO Regio Arnhem-Nijmegen)
Record Dates: First submitted 2021-07-28; First posted 2021-08-11 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer Metastatic; Prostate Cancer; Lymph Node Metastases
MeSH Terms: conditions — Prostatic Neoplasms; Lymphatic Metastasis | interventions — Nomograms

STUDY DESIGN:
Intervention Model Description: Intervention
  PSMA PET/CT based indication for ePLND:
  1. Node-negative PSMA PET/CT [N0] and M0: do not perform ePLND
  2. Node-positive PSMA PET/CT [N1] and M0: perform ePLND
  Comparator Nomogram-based indication for ePLND (conform current EAU guidelines)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PSMA PET/CT based indication for ePLND: (Experimental): 1. Node-negative PSMA PET/CT [N0] and M0: do not perform ePLND
  2. Node-positive PSMA PET/CT [N1] and M0: perform ePLND
  Interventions: Device: PSMA-PET/CT
- Nomogram-based indication for ePLND (standard of care) (Active Comparator): Nomogram-based indication for ePLND (conform current EAU guidelines)
  Interventions: Other: Nomogram

INTERVENTIONS:
Device: PSMA-PET/CT — In the intervention arm patients will only undergo ePLND in addition to robot-assisted radical prostatectomy (RARP) in case of suspected LNI on PSMA PET/CT (miN1), whereas ePLND will be omitted in those without PSMA positive lymph nodes (miN0).
  Arms: PSMA PET/CT based indication for ePLND:
Other: Nomogram — Current standard of care includes performing extended pelvic lymph node dissection (ePLND) in all patients with primary prostate cancer and a nomogram-based risk of LNI >5%
  Arms: Nomogram-based indication for ePLND (standard of care)

SUMMARY:
To determine if the use of Prostate-Specific Membrane Antigen Positron Emission Computer Tomography (PSMA PET/CT) as a selection tool for performing extended lymph node dissection (ePLND) for prostate cancer (PCa) in the primary staging setting results in fewer ePLND procedures and therefore lower overall healthcare costs, lower patient burden in terms of intervention-related complications and morbidity, with comparable disease prognosis, compared to the current European Guideline-recommended standard practice which includes performing ePLND in PCa patients who are candidates for active treatment with a nomogram-calculated lymph node involvement (LNI) risk >5%.

DETAILED DESCRIPTION:
Background: Use of prostate-specific membrane antigen (PSMA) positron emission tomography (PET) - computer tomography (CT) has drastically improved the ability to detect and exclude presence of pelvic lymph node invasion (LNI) compared to conventional imaging. However, current standard of care still includes performing extended pelvic lymph node dissection (ePLND) in all patients with primary prostate cancer and a nomogram-based risk of LNI >5%. It is unclear if use of PSMA PET/CT as a triage test can safely reduce the number of ePLND and hence reduce the associated morbidity and costs, without negatively influencing disease prognosis.

Objective: To assess whether PSMA PET/CT can be safely used as a triage test for selecting primary prostate cancer patients for ePLND. We will additionally assess cost-effectiveness of the PSMA PET/ CT triage strategy.

Design, setting and Participants: THE PSMA-SELECT trial includes patients with biopsy-confirmed prostate cancer, without evidence of distant metastasis (M0) on PSMA PET/CT, opting for treatment with radical prostatectomy (RP), with a nomogram-calculated risk of LNI >5%. Patients will be randomized 1:1. In the intervention arm patients will only undergo ePLND in addition to robot-assisted radical prostatectomy (RARP) in case of suspected LNI on PSMA PET/CT (miN1), whereas ePLND will be omitted in those without PSMA positive lymph nodes (miN0). In the control arm, all patients will undergo ePLND in addition to RARP.

Outcome measurements and statistical analysis: The primary endpoint of this study is biochemical recurrence rate at two years post-surgery. Secondary outcome measures are number of ePLNDs indicated and performed, treatment-related adverse events, initiation of salvage treatment, metastasis-free survival, patient-reported outcome measures and individual and cumulative healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the prostate
* Indication for ePLND combined with robot assisted radical prostatectomy (RARP) (MSKCC nomogram >5%, if not applicable when only MRI targeted biopsies are positive, the Briganti nomogram will be used)
* Suitable for robot-assisted ePLND and RARP
* Mentally competent and understanding of benefits and potential burden of the study
* Written informed consent
* No known allergies for PSMA tracer.

Exclusion Criteria:

* History of prior diagnosed or treated PCa
* Known concomitant malignancies (except Basal Cell Carcinoma of the skin)
* Unwillingness or inability to undergo PSMA PET/CT and/or ePLND and RARP
* PSMA non-avid PCa (local tumor activity)
* Presence of distant metastasis (M1)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference in biochemical recurrence rate between groups. | 2 years
  Biochemical recurrence (BCR) is defined as the occurrence of measurable (>0.2 ng/ml) prostate specific antigen (PSA), during routinely follow-up up to five years after surgery, determined at two different occasions with at least one week between them.The BCR-rate between the control group and intervention groups will be compared.

SECONDARY OUTCOMES:
Total number of ePLNDs and PSMA PET/CTs performed and their intervention-related healthcare costs | up to 5 years post-surgery
  Total number of ePLNDs and PSMA PET/CTs performed and their intervention-related healthcare costs such as consumption of operation room (OR) time, costs of complication-related interventions and associated (prolonged) hospital stay.
Incidence and types of surgical complications after RARP and ePLND | up to 1 year post-surgery
  Surgical complications are graded according to the Clavien-Dindo Classification, defined as:
  Grade 1 = Any deviation from the normal postoperative course. Grade 2 = Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Grade 3 = Requiring surgical, endoscopic or radiological intervention, not under (Grade 3a) or under general anesthesia (Grade 3b). Grade 4 = Life-threatening complication with single organ (Grade 4a) or Multiorgan dysfunction (Grade 4b). Grade 5 = Death of a patient.
Total nodes resected on ePLND and number of positive and negative nodes within and outside of the standard ePLND template | up to 5 years post-surgery
  Total nodes resected on ePLND and number of positive and negative nodes within and outside of the standard ePLND template as described by the EAU guidelines.
Occurrence of pelvic lymph node metastasis and distant metastasis (visceral, bone, distant lymph nodes, pelvic lymph nodes) on PSMA-PET/CT during follow-up | up to 5 years post-surgery
  Time to appearance of pelvic lymph node metastasis (N1) and distant metastasis (M1) using PSMA PET/CT
Initiation of salvage therapy | up to 5 years post-surgery
  The time from surgery to the start of salvage therapy (salvage ePLND, salvage radiation treatment, systemic treatment [androgen deprivation therapy (ADT) and eventual additional chemotherapy]).
Metastasis-free survival | up to 5 years post-surgery
  The time from surgery to the time of the scan that showed first evidence of radiographically detected bone or soft tissue distant metastasis.
Hormone-therapy free survival | up to 5 years post-surgery
  The time from surgery to the start of hormone therapy (ADT)
Diagnostic accuracy measures of PSMA PET/CT | up to 5 years post-surgery
  Diagnostic accuracy measures including per-patient and per-template sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of PSMA PET/CT for the detection of lymph node metastasis at baseline and, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60 months post-surgery.
(Changes) in the EPIC-26 sexual functioning domain score between groups | up to 5 years post-surgery
  Expanded Prostate Cancer Index Composite (EPIC)-26 will be used to measure sexual functioning. EPIC-26 contains five symptom domains (urinary incontinence, urinary irritative/obstructive, sexual, bowel, hormonal), scored from 0 (worst) to 100 (best). Questionnaires will be send out at baseline (diagnosis) and 12, 24, 36, 48 and 60 months following surgery.
(Changes in) quality-adjusted life-years (EQ-5D-5L) in patients in the control group vs. intervention group | up to 5 years post-surgery
  The EuroQol (EQ)-5 Dimension (D)-5 Level (L) is a health-related quality of life questionnaire which can be used to derive utilities from patients. The EQ-5D-5L descriptive system comprises five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety. Each domain has 5 response levels: (1) no problems, (2) slight problems (3) moderate problems (4) severe problems and (5) unable to/extreme problems.
  Questionnaires will be administered at baseline, 12, 24, 36, 48 and 60 months following diagnosis.
Total health care related costs (iMTA MCQ) in patients in the control group vs. intervention group | up to 5 years post-surgery
  The institute for Medical Technology Assessment (iMTA) Medical Consumption Questionnaire (MCQ) measures all relevant health care related costs. The iMCQ includes questions related to frequently occurring contacts with health care providers. Questionnaires will be send out at baseline and 3, 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60 months post-surgery.
Total loss of productivity and presenteeism (iMTA PCQ) in patients in the control group vs. intervention group | up to 5 years post-surgery
  The institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire (PCQ) measures loss of productivity due to illness or recovery in patients below the age of 65 years based on patient reported absences from paid (or unpaid) labor. Questionnaires will be send out to each individual patient at baseline and, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul A. van Basten, Principal Investigator — Canisius-Wilhelmina Hospital
Locations (1):
- Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided